CLINICAL TRIAL: NCT06029517
Title: A Novel Sugar-Sweetened Beverage Reduction Intervention for Native American Men
Brief Title: A Sugar-Sweetened Beverage Reduction Intervention for Native American Men
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: I 810620; R56NR019498 (NIH)
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Cardiovascular Disorder; Coronary Artery Disease; Diabetes Mellitus; Obesity-Related Malignant Neoplasm
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease; Diabetes Mellitus | interventions — Early Intervention, Educational; Educational Status; Methods; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aim 1 - interview, focus group (Other): Participants complete interviews over 60 minutes and attend focus groups over 90 minutes in support of intervention adaptation and refinement
  Interventions: Other: Interview; Procedure: Discussion
- Aim 2 - Indigenous SIPin (Experimental): Participants receive the Indigenous SIPin intervention over 6 months, which includes in-person and/or virtual educational sessions weekly over 30 minutes for 12 weeks and text message communications BIW for 12 weeks and then monthly thereafter up to month 6.
  Interventions: Other: Education Intervention

INTERVENTIONS:
Other: Education Intervention — Receive Indigneous SIPin intervention
  Other Names: Education for Intervention
  Arms: Aim 2 - Indigenous SIPin
Other: Interview — Complete interviews
  Arms: Aim 1 - interview, focus group
Procedure: Discussion — Attend focus groups
  Arms: Aim 1 - interview, focus group

SUMMARY:
This clinical trial develops and tests a culturally-appropriate educational program (Indigenous SIPin) for reducing sugar-sweetened beverage consumption in men affiliated with Native American athletics communities. Sugary drinks are drinks like pop, soda, and juice. Increased sugar consumption may lead to an increased risk of chronic diseases, including obesity, diabetes, some types of obesity-related cancers, coronary heart disease, hypertension, and dental decay. A culturally sensitive program may help reduce sugar-sweetened beverage consumption in Native American men

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Conduct and analyze qualitative data from focus groups and key informant interviews with Native American community members including Native American leaders and community members to develop Sugar Sweetened Beverage (SSB) intervention for Native American men (SIPsmartER Lacrosse).

OUTLINE:

AIM 1: Participants complete interviews over 60 minutes and attend focus groups over 90 minutes in support of intervention adaptation and refinement.

AIM 2: Participants receive the Indigenous SIPin intervention over 6 months, which includes in-person and/or virtual educational sessions weekly over 30 minutes for 12 weeks and text message communications twice a week (BIW) for 12 weeks and then monthly thereafter up to month 6.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years or older
* Research conducted on tribal lands require tribal government approval. Our project will not be occurring on tribal lands. The project will be working with Native organizations off-territory
* Participants only must own a smart device in order to receive study text messages
* At least 18 years or older
* Research conducted on tribal lands require tribal government approval. Our project will not be occurring on tribal lands. The project will be working with Native organizations off-territory
* Participants only must own a smart device in order to receive study text messages

Exclusion Criteria:

* Research conducted on tribal lands require tribal government approval. Since we do not currently have tribal government approval, our project will not be occurring on tribal lands

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in SSB intake for men affiliated with Native American athletic communities | up to 6 months
  Will conduct half hour classes with the Native American community members on how to improve wellness and drink less sugary drinks

SECONDARY OUTCOMES:
Sugar sweetened beverage intake | Baseline to 6 months
  change in consumption of sugar sweetened beverages
Change in body weight | baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rodney Haring, Principal Investigator — Roswell Park
Locations (1):
- Roswell Park Comprehensive Cancer Center, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2023-07-07): https://cdn.clinicaltrials.gov/large-docs/17/NCT06029517/ICF_000.pdf